CLINICAL TRIAL: NCT03164213
Title: Facilitation of Brain Plasticity for Language Recovery in Patients With Aphasia Due to Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nachum Soroker, MD (Other)
Responsible Party: Sponsor-Investigator, Nachum Soroker, MD, Head, Department of neurologic rehabilitation, Loewenstein, Loewenstein Hospital
Organization: Loewenstein Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: loe170037ctil
Record Dates: First submitted 2017-04-24; First posted 2017-05-23 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Stroke; Aphasia
Keywords: tDCS; aphasia
MeSH Terms: conditions — Stroke; Aphasia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental tDCS (Experimental): TDCS stimulation at the left M1 region followed by naming therapy. The intervention will be given daily for duration of two weeks (5 days/week).
  Interventions: Device: experimental: tDCS
- sham tDCS (Sham Comparator): Sham tDCS at the left M1 region followed by naming therapy. The intervention will be given daily for duration of two weeks (5 days/week).
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: experimental: tDCS — The anode will be placed over the left M1 representation of the hand (C3 of the 10-20 EEG system). Twenty minutes of anodal-tDCS (1mA) will be administered at the beginning of the daily treatment session. Following the stimulation will be 45 minutes of naming therapy.
  Other Names: tDCS
  Arms: Experimental tDCS
Device: sham tDCS — The anode will be placed over the left M1 representation of the hand (C3 of the 10-20 EEG system). Twenty minutes of sham-tDCS will be administered at the beginning of the daily treatment session.
  During sham-tDCS, the current will be ramped up and remained at 1mA only for 30 s before ramping down, which does not affect neural functions, but assures effective blinding of participants due to the initial tingling sensation on the scalp. Following the sham stimulation will be 45 minutes of naming therapy.
  Arms: sham tDCS

SUMMARY:
The purpose of this study is to investigate effects of tDCS stimulation in the left primary motor area followed by naming therapy to improve language functions in patients with aphasia in the sub-acute stage.

DETAILED DESCRIPTION:
Transcranial Direct Current Stimulation (tDCS) is a simple and non-intrusive method that has demonstrated promising results in language rehabilitation of patients with aphasia. Various studies have used different stimulation set-ups, some based on prior structural and functional brain mapping in order to choose the optimal stimulation region. An additional approach that was found beneficial is stimulation of the left primary motor area (M1). A major advantage of this approach is its relative simplicity that may increase the application of this intervention in clinical settings. This intervention approach has been studied in patients with chronic aphasia and targeted on naming ability. In the current study the investigators aim to study the influence of a stimulation set-up at M1 in stroke patients suffering from aphasia that are in the sub-acute stage. In addition the investigators aim to study additional language functions including pragmatics and grammar. The study will include 30 patients suffering from aphasia which are in the sub-acute stage. The patients will undergo complete language assessments at 3 time points: baseline, post intervention (third week from recruitment) and one month follow-up. The study group will include 15 patients that will undergo TDCS at the left M1 region followed by naming therapy. The intervention will be given daily for duration of two weeks (5 days/week). The control group will include 15 patients that will undergo the same protocol apart from sham TDCS. The effect of the intervention will be examined taking into account the extent and location of the brain damage on language functions.

ELIGIBILITY:
Inclusion Criteria:

* patients post stroke with right hemiplegia and aphasia with cognitive capacity to understand instructions and at the aphasia cut-of level defined by "SHEMESH" assessment

Exclusion Criteria:

* unstable clinical state, craniotomy, epilepsy, heart pacer or lack of cooperation

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in "Shemesh" 100 nouns test (Biran and Friedmann 2005) | baseline (before intervention), post intervention (on the third week from recruitment) and one month follow-up.
  language test

SECONDARY OUTCOMES:
Change in Western Aphasia Battery Hebrew | baseline (before intervention), post intervention (on the third week from recruitment) and one month follow-up.
  aphasia assessment
Change in Psycholinguistic Assessments of Language Processing in Aphasia | baseline (before intervention), post intervention (on the third week from recruitment) and one month follow-up.
  psycholinguistical assessment of aphasia

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Soroker, M.D., Principal Investigator — Loewenstein Hospital